CLINICAL TRIAL: NCT03435185
Title: Greater Occipital and Supraorbital Nerve Blockade For The Preventive Treatment of Migraine
Brief Title: Greater Occipital and Supraorbital Nerve Blockade in Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cem Bölük, Medical Doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/514/85/5
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Results first posted 2019-07-22 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Migraine Disorders
Keywords: Pain; Nerve Blocks; Headache; Local Anaesthetics; Migraine
MeSH Terms: conditions — Migraine Disorders; Pain; Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blockade Group (Active Comparator): Lidocaine injections. Procedure. Grater occipital nerve and supraorbital nerve were blocked with %2 lidocaine. These injections were repeated weekly for three weeks. After treatment was completed, patients were followed up for 2 months at the polyclinic to assess the clinical response.
  Interventions: Procedure: Lidocaine injections
- Placebo Group (Placebo Comparator): Saline injections. Procedure. Grater occipital nerve and supraorbital nerve were injected with saline.These injections were repeated weekly for three weeks. After treatment was completed, patients were followed up for 2 months at the polyclinic to assess the clinical response.
  Interventions: Procedure: Saline injections

INTERVENTIONS:
Procedure: Lidocaine injections — Lidocaine injections. A mixture of 1 ml 2% lidocaine and 0.9% 1 ml saline was injected bilaterally to greater occipital nerve and supraorbital nerve in the blockade patients.
  Arms: Blockade Group
Procedure: Saline injections — Saline injections. Patients received 2 ml 0.9% saline in bilaterally to greater occipital nerve and supraorbital nerve
  Arms: Placebo Group

SUMMARY:
The investigators aimed to evaluate the efficacy of greater occipital nerve and supraorbital nerve blockade with local anesthetics for the preventive treatment of migraine without aura.

DETAILED DESCRIPTION:
A mixture of 1 ml 2% lidocaine and 0.9% 1 ml saline was injected bilaterally to GON and SON in the blockade patients. Placebo patients received 2 ml 0.9% saline in the same way. Patients were blinded to kind of injection.

ELIGIBILITY:
Inclusion Criteria:

* Lack of benefits 1 year from preventive treatment or intolerance to their treatments.
* 18 ≥ years old
* Migraine without aura for more than 1 year, minimum of two or more migraine attacks per month.

Exclusion Criteria:

* Patients with any chronic illness, medication overuse headache, a history of cranial and cervical surgery
* Allergies to local anesthetics
* Hemorrhagic diathesis
* Alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2016-06-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang Y, Kang J, Zhang Y, Zhang X. Influence of greater occipital nerve block on pain severity in migraine patients: A systematic review and meta-analysis. Am J Emerg Med. 2017 Nov;35(11):1750-1754. doi: 10.1016/j.ajem.2017.08.027. Epub 2017 Aug 14. PMID 28844531

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 patients were excluded due to not meeting inclusion criteria
Groups:
- Blockade Group: Grater occipital nerve and supraorbital nerve blockade injections with %2 lidocaine
  Lidocaine injections: Lidocaine injections. A mixture of 1 ml 2% lidocaine and 0.9% 1 ml saline was injected bilaterally to greater occipital nerve and supraorbital nerve in the blockade patients.
- Placebo Group: Grater occipital nerve and supraorbital nerve injections with saline
  Saline injections: Saline injections. Patients received 2 ml 0.9% saline in bilaterally to greater occipital nerve and supraorbital nerve
Period: Overall Study
Arm/Group | Blockade Group | Placebo Group
Started | 44 | 43
Completed | 43 | 28
Not Completed | 1 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blockade Group | Placebo Group | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 43 | 87
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change of Frequency of Headache
Description: Number of headache days in a month. Scores from both months were averaged. Minimum=0 Maximum=30. Lower scores mean a better outcome.
Time Frame: Patients were followed up from baseline to 2 months after first injection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blockade Group | Placebo Group
Number analyzed (Participants) | 43 | 28
score on a scale | 5.3 (7.4) | 7.5 (7.2)

2. Primary Outcome: Change of Severity of Headache
Description: Mean visual analog scale (VAS) scores. Scores from both months were avareged. Minimum=0 Maximum=10. Lower scores mean a better outcome
Time Frame: Patients were followed up for 2 months from baseline after first injection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blockade Group | Placebo Group
Number analyzed (Participants) | 43 | 28
score on a scale | 5.5 (1.9) | 7.4 (1.3)

ADVERSE EVENTS:
Time Frame: 10 months
Description: Clinically observed adverse events
Arm/Group | Blockade Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/28
Other Adverse Events (participants affected / at risk) | 37/43 | 19/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blockade Group (N=43) | Placebo Group (N=28)
Minor Bleedings (Skin and subcutaneous tissue disorders) | 37 | 19 — Minor bleedings due to injections

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes